CLINICAL TRIAL: NCT06474663
Title: A Phase I Study Investigating the Combination of Cladribine, Low Dose Cytarabine and Sorafenib Alternating With Decitabine in Pediatric Relapsed and Refractory Acute Leukemias
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: 0 participants
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0302; NCI-2024-05386 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Refractory Acute Leukemia; Relapsed Acute Leukemia
MeSH Terms: interventions — Cladribine; Cytarabine; Sorafenib; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 (Experimental): Participants enrolled in Phase 1, the dose level of cladribine, cytarabine, decitabine, and sorafenib will depend on when you join this study. Up to 2 dose levels of this drug combination may be tested. Between 3-6 participants will be enrolled in each dose level. The first group of participants will receive the starting dose level of this drug combination. If no intolerable side effects are seen, the next group of participants will receive the higher dose level of this drug combination.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: Sorafenib; Drug: Decitabine
- Dose Expansion (Experimental): Participants enrolled in Dose Expansion, you will receive cladribine, cytarabine, decitabine, and sorafenib at the recommended dose level found in Phase 1.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: Sorafenib; Drug: Decitabine

INTERVENTIONS:
Drug: Cladribine — Given by IV
  Other Names: Leustatin®; 2-CdA
Drug: Cytarabine — Given by SC
  Other Names: Ara-C; Cytosar®; DepoCyt™; Cytosine arabinosine hydrochloride
Drug: Sorafenib — Given by PO
  Other Names: Nexavar®; BAY 43-9006
Drug: Decitabine — Given by IV

SUMMARY:
To find the recommended dose of the drug combination cladribine, cytarabine, decitabine, and sorafenib in participants with relapsed/refractory AML, MPAL, and ALAL.

DETAILED DESCRIPTION:
Primary Objectives - To determine the safety, tolerability, and recommended phase II dose (RP2D) of the combination of cladribine, low-dose cytarabine, sorafeneib alternating with decitabine for pediatric participants with acute leukemias.

Secondary Objectives

- To determine the preliminary assessment of efficacy by overall response (OR), including complete remission (CR), CR with partial hematological recovery (CRh), CR with incomplete blood count recovery (CRi), Morphologic leukemia free state (MLFS) and partial remission (PR), overall survival (OS), event-free survival (EFS) and duration of response (DOR) of pediatric participants treated with this combination.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 1 year to 21 years
2. ECOG performance status of ≥ 2.
3. Relapsed21/refractory: AML22 or Mixed phenotype acute leukemia (MPAL) patients /Acute leukemia of ambiguous lineage (ALAL) with.

   1. ≥1% leukemic blasts in the bone marrow:
   2. As detected by MRD testing ≥ 25% or MRD is ≥ 5% with 1 additional sensitive diagnostic test demonstrating .1% blasts (NGS-MRD (clonoSeq23) or FISH or cytogenetics or RT-PCR of leukemic specific marker or M2/M3 morphology); or MRD is ≥ 1% with 2 additional sensitive diagnostic tests demonstrating ≥1% blasts.

   i. If the MRD is ≥ 1% but without the required confirmatory tests, then a relapse can still be defined if a consecutive marrow evaluation separated by ≥1 week demonstrates. ≥ 1% using 2 sensitive diagnostic tests.

   ii. If MRD testing is unavailable, then a single marrow is sufficient to define relapse if M3 morphology or M2 morphology with 1 additional sensitive diagnostic test demonstrating ≥1% blasts (FISH or cytogenetics or RT-PCR of leukemic specific marker) or M1 morphology with 2 additional sensitive diagnostic tests demonstrating. ≥1% blasts is present.

   iii. If the morphology is M2 with no confirmatory tests, then a relapse can still be defined if a consecutive marrow evaluation separated by ≥ 1 week demonstrates M2 morphology.

   c. Marrow definitions: M2 marrow ≥ 5 to <25% blasts; M3 marrow ≥ 25% blasts
4. WBC must be below 25,000/ ƒÊL at time of enrollment. Patients may receive cytoreduction prior to enrollment.
5. Baseline ejection fraction must be > 40%.
6. Adequate hepatic function (direct bilirubin < 1.5x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement, and AST and/or ALT < 5x ULN unless considered due to leukemic involvement, in which case direct bilirubin or AST and/or ALT < 5x ULN will be considered eligible).
7. Adequate renal function (creatinine clearance ≥ 30 mL/min) unless related to disease. (Justification on page 7-8)
8. In the absence of rapidly proliferative disease, the interval from prior treatment to time of initiation will be at least 14 days for cytotoxic or non-cytotoxic (immunotherapy agent(s), or an interval of 5 half-lives of the prior therapy. Oral hydroxyurea and/or cytarabine (up to 2 g/m2) for patients with rapidly proliferative disease is allowed before the start of study therapy, as needed, for clinical benefit and after discussion with the PI. Concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted.
9. Unless surgically or biologically sterile: Women of childbearing potential must agree to adequate methods of contraception during the study and at least 3 months for males, and 6 months for females, after the last treatment.

Exclusion Criteria:

1. Participants who weigh less than 10kg.
2. Participants with any concurrent uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place the participant at unacceptable risk of study treatment.
3. The use of other chemotherapeutic agents or anti-leukemic agents is not permitted during study with the following exceptions (1) intrathecal chemotherapy for prophylactic use or for controlled CNS leukemia. (2) use of hydroxyurea for patients with rapidly proliferative disease or for control of counts during differentiation syndrome. (3) use of steroids for treatment of differentiation syndrome.
4. Participants with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications.
5. Participants with a concurrent active malignancy under treatment.
6. Known active hepatitis B (HBV) or Hepatitis C (HCV) infection or known HIV infection.
7. Female participants who are pregnant or breast-feeding.
8. Participants has an active uncontrolled infection.
9. History of or any concurrent condition, therapy, or laboratory abnormality that in the Investigator's opinion might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the participants.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-31 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Branko Cuglievan, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org